CLINICAL TRIAL: NCT06127641
Title: Rehabilitation of People With Post-tuberculosis Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 70493823.5.0000.5259
Record Dates: First submitted 2023-10-29; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Tuberculosis
Keywords: Pulmonary tuberculosis; Tuberculosis sequelae; Rehabilitation; ADL-Glittre test; Functionality; Quality of life
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants will receive standard care (SC)
  Interventions: Other: Standard Care
- Intervention (Experimental): Participants will receive the standard care (SC) plus pulmonary rehabilitation (PR)
  Interventions: Other: Standard care plus pulmonary rehabilitation

INTERVENTIONS:
Other: Standard care plus pulmonary rehabilitation — A 12-week rehabilitation program, 3X/week. Each outpatient session will last 2 hours including: guidance on the care of inhalation techniques and/or oxygen therapy, when prescribed; aerobic training on a cycle ergometer supervised by a physiotherapist (30 min each: 5 min warm-up, 20 min training and 5 min cool-down) at constant load calculated with Hill's equation (HILL et al., 2008). Optional components of RP will include: inspiratory muscle conditioning using a threshold-loading device, inspiratory muscle training with powerbreathe, breathing exercises, airway clearance, psychological support, relaxation and nutritional counseling. Patients will participate in two group educational sessions, managed by a respiratory physiotherapist, on lifestyle, physical activity and maintenance programs (VISCA et al., 2019; FUGAZZARO et al., 2017; TENCONI et al., 2021).
  Arms: Intervention
Other: Standard Care — Participants will receive standard care (SC): a therapeutic education session upon admission, as well as pulmonary rehabilitation (PR) taught by a physical therapist. This therapeutic educational session will involve counseling and self-care management, emphasizing breathing exercises and sputum clearance and self-care techniques. It will consist of smoking cessation education (if this is the case, as tobacco is associated with TB), respiratory retraining (pursed lip breathing, diaphragmatic breathing and segmental breathing) and secretion removal training (coughing exercise, huffing , assisted cough and postural drainage).
  Arms: Control

SUMMARY:
Tuberculosis (TB) can leave numerous sequelae, where survivors experience a transition from an acute illness to living with a multifaceted chronic illness. Post-TB lung disease (PD-PTB) encompasses lung diseases and pathologies that occur after one or more episodes of TB, which can affect the patient's lung health and cause disabling symptoms that strongly affect their long-term health. In 2020, it was estimated that there were 155 million TB survivors still alive worldwide, with a large proportion of them carrying functional sequelae with profound socioeconomic repercussions. Thus, the aim of this study is to evaluate the effect of pulmonary rehabilitation (PR) on functionality and health-related quality of life (HRQoL) of people with PD-PTB and to build a PD-PTB severity scoring system based on the data. of pre-RP individuals using artificial intelligence technique.

DETAILED DESCRIPTION:
Tuberculosis (TB) can leave numerous sequelae, where survivors experience a transition from an acute illness to living with a multifaceted chronic illness. Post-TB lung disease (PD-PTB) encompasses lung diseases and pathologies that occur after one or more episodes of TB, which can affect the patient's lung health and cause disabling symptoms that strongly affect their long-term health. In 2020, it was estimated that there were 155 million TB survivors still alive worldwide, with a large proportion of them carrying functional sequelae with profound socioeconomic repercussions. Thus, the aim of this study is to evaluate the effect of pulmonary rehabilitation (PR) on functionality and health-related quality of life (HRQoL) of people with PD-PTB and to build a PD-PTB severity scoring system based on the data. of pre-RP individuals using artificial intelligence technique. This is a randomized controlled trial, in which the sample will be divided into two groups: intervention for 12 weeks with PR and standard care. Functional capacity will be evaluated pre- and post-PR through the Glittre-ADL test with incorporation of dynamic ventilation, lung function (including impulse oscillometry), respiratory and peripheral muscle function, general fatigue and HRQoL. It is expected that PTB-PD patients will benefit significantly and, therefore, be able to (re)enter society, especially in job market.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-tuberculosis lung disease, clinically stable and able to perform >80% of training sessions.

Exclusion Criteria:

* Presence of comorbidities not related to PD-PTB.
* Patients with inability to perform TGlittre.
* Patients who have cognitive changes that impair their inclusion in the study.
* Treatment abandonment during the application of the PR protocol.
* Uncontrolled hypertension or use of psychotropic medications.
* Any significant limitations due to osteoarthropathy.
* Having had any orthopedic surgery in the previous year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional capacity using the ADL-Glittre test (TGlittre) incorporated into dynamic ventilation before and after the PR program | an average of 4 years
  Executed as proposed by Skumlien et al. (2006). The shorter duration TGlittre will be used for analysis and comparison to predicted values for healthy brazilians (REIS et al., 2018). Furthermore, the device Spiropalm 6MWT, Cosmed, Rome, Italy, will be attached to the patient. Inspiratory capacity (IC) will be obtained before and after TGlittre, and a ≥100 mL decrease in IC (∆IC) during exertion will be defined as dynamic hyperinflation (TOSUN et al., 2022). Other dynamic ventilatory responses assessed: minute ventilation (VE) and ventilatory reserve (RV). The latter indicates how close VE comes to maximum ventilation during a given activity, and will be calculated as the difference between maximum voluntary ventilation (MVV) and VEpeak ([MVV - VEpeak]/VVM); VR <30% will be considered exertional ventilation limitation (LOPES et al., 2011a). The MVV will be automatically determined by the device as 40 multiplied by FEV1

SECONDARY OUTCOMES:
Clinical-functional assessment | an average of 4 years
  Clinical examination and anthropometric measurements
Saint George's Respiratory Questionnaire (SGRQ) | an average of 4 years
  To measure health-related quality of life (HRQOL), the SGRQ will be applied, which was previously validated and adapted for the Brazilian population (DE SOUSA et al., 2000). This instrument covers aspects in 3 domains, which are: symptoms, activity and psychosocial impacts that the disease can influence on your daily routine. The answers translate into points that, once added together, can infer an altered HRQoL in a given domain.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | an average of 4 years
  The FACIT-F was translated into Portuguese by the FACIT.ORG group. It is a 13-item scale that aims to assess the individual's general fatigue correlated to their daily activities. These items provide a score ranging from 0 to 52. The lower the score, the lower the fatigue index. A score greater than 30 indicates severe fatigue. Clinically, an increase of 3 to 4 points in FACIT-F is considered an important difference (MIYAMOTO, 2016; LIMA et al., 2019).
Pulmonary function measurements | an average of 4 years
  Pulmonary function using an HDpft 3000 device (nSpire Health, Inc., Longmont, CO, USA). Spirometry, body plethysmography, carbon monoxide diffusion (DLCO) measurement and respiratory muscle strength measurement will be performed.
Handgrip strength (HGS) | an average of 4 years
  HGS will be measured in kilograms using a digital dynamometer (SH5001, Saehan Corporation, Korea). HGS will be assessed with participants sitting in an armless chair, with elbow flexion at 90°, forearms in a neutral position and wrist extension between 0 and 30° (NONATO et al., 2020). Maximum strength will be assessed after a sustained contraction of 3 s in the dominant hand; the highest value of 3 attempts with 1 min intervals will be considered for analysis (ASSIS et al., 2022)
Quadriceps strength (QS) | an average of 4 years
  QS will be evaluated using a traction dynamometer with a sensor capacity of 200 kg (E-lastic 5.0, E-sporte SE, Brazil). The range of movement when performing the test will be determined at 90°, starting from 90° with the knee in flexion. Maximum strength will be assessed after a sustained contraction of 5 s in the dominant leg, with the highest value of 3 attempts at 1 min intervals being considered for analysis (ASSIS et al., 2022).

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Agnaldo José Lopes, Rio de Janeiro
  - Centro Universitario Augusto Motta, Rio de Janeiro

REFERENCES:
- [Background] Aggarwal AN, Gupta D, Janmeja AK, Jindal SK. Assessment of health-related quality of life in patients with pulmonary tuberculosis under programme conditions. Int J Tuberc Lung Dis. 2013 Jul;17(7):947-53. doi: 10.5588/ijtld.12.0299. PMID 23743314
- [Background] Allwood BW, van der Zalm MM, Amaral AFS, Byrne A, Datta S, Egere U, Evans CA, Evans D, Gray DM, Hoddinott G, Ivanova O, Jones R, Makanda G, Marx FM, Meghji J, Mpagama S, Pasipanodya JG, Rachow A, Schoeman I, Shaw J, Stek C, van Kampen S, von Delft D, Walker NF, Wallis RS, Mortimer K. Post-tuberculosis lung health: perspectives from the First International Symposium. Int J Tuberc Lung Dis. 2020 Aug 1;24(8):820-828. doi: 10.5588/ijtld.20.0067. PMID 32912387
- [Background] Allwood BW, Maasdorp E, Kim GJ, Cooper CB, Goldin J, van Zyl-Smit RN, Bateman ED, Dawson R. Transition from Restrictive to Obstructive Lung Function Impairment During Treatment and Follow-Up of Active Tuberculosis. Int J Chron Obstruct Pulmon Dis. 2020 May 11;15:1039-1047. doi: 10.2147/COPD.S219731. eCollection 2020. PMID 32494129
- [Background] Amaral AF, Coton S, Kato B, Tan WC, Studnicka M, Janson C, Gislason T, Mannino D, Bateman ED, Buist S, Burney PG; BOLD Collaborative Research Group. Tuberculosis associates with both airflow obstruction and low lung function: BOLD results. Eur Respir J. 2015 Oct;46(4):1104-12. doi: 10.1183/13993003.02325-2014. Epub 2015 Jun 25. PMID 26113680
- [Background] Banu Rekha VV, Ramachandran R, Kuppu Rao KV, Rahman F, Adhilakshmi AR, Kalaiselvi D, Murugesan P, Sundaram V, Narayanan PR. Assessment of long term status of sputum positive pulmonary TB patients successfully treated with short course chemotherapy. Indian J Tuberc. 2009 Jul;56(3):132-40. PMID 20349754
- [Background] Bogossian M, Santoro IL, Jamnik S, Romaldini H. Bronchiectasis: a study of 314 cases tuberculosis x nontuberculosis. J Bra Pneumol. 1998; 24(1): 11-6.
- [Background] Brasil. Ministério da Saúde. Manual de Recomendações para o Controle da Tuberculose no Brasil 2019. Disponível em: https://bvsms.saude.gov.br/bvs/publicacoes/manual_recomendacoes_controle_tuberculose_brasil_2_ed.pdf
- [Background] Butzko RP, Sotolongo AM, Helmer DA, Klein-Adams JC, Osinubi OY, Berman AR, Ortiz-Pacheco R, Falvo MJ. Forced oscillation technique in veterans with preserved spirometry and chronic respiratory symptoms. Respir Physiol Neurobiol. 2019 Feb;260:8-16. doi: 10.1016/j.resp.2018.11.012. Epub 2018 Nov 30. PMID 30508589
- [Background] Byrne AL, Marais BJ, Mitnick CD, Lecca L, Marks GB. Tuberculosis and chronic respiratory disease: a systematic review. Int J Infect Dis. 2015 Mar;32:138-46. doi: 10.1016/j.ijid.2014.12.016. PMID 25809770
- [Background] Chin AT, Rylance J, Makumbirofa S, Meffert S, Vu T, Clayton J, Mason P, Woodruff P, Metcalfe J. Chronic lung disease in adult recurrent tuberculosis survivors in Zimbabwe: a cohort study. Int J Tuberc Lung Dis. 2019 Feb 1;23(2):203-211. doi: 10.5588/ijtld.18.0313. PMID 30808453
- [Background] Daniels KJ, Irusen E, Pharaoh H, Hanekom S. Post-tuberculosis health-related quality of life, lung function and exercise capacity in a cured pulmonary tuberculosis population in the Breede Valley District, South Africa. S Afr J Physiother. 2019 Jul 31;75(1):1319. doi: 10.4102/sajp.v75i1.1319. eCollection 2019. PMID 31392293
- [Background] De Sousa TC, Jardim JR, Jones P. Validation of the Saint George's Respiratory Questionnaire in patients with chronic obstructive pulmonary disease in Brazil. J Pneumologia 2000; 26(3): 119-128.
- [Background] Dias VL, Canan MGM, Leitao CA, Okuno EA, de Sant'Ana GRD, Miranda JV. Profile of patients with post-tuberculosis bronchiectasis in a tertiary care hospital in Brazil. J Clin Tuberc Other Mycobact Dis. 2022 Nov 13;29:100339. doi: 10.1016/j.jctube.2022.100339. eCollection 2022 Dec. PMID 36405996
- [Background] Ehrlich RI, White N, Norman R, Laubscher R, Steyn K, Lombard C, Bradshaw D. Predictors of chronic bronchitis in South African adults. Int J Tuberc Lung Dis. 2004 Mar;8(3):369-76. PMID 15139477
- [Background] Evans D. Socio-economic consequences and quality adjusted life years associated with post-TB sequelae. Int J Tuberc Lung Dis. 2021; 25(Suppl 2): S21.
- [Background] Fugazzaro S, Costi S, Mainini C, Kopliku B, Rapicetta C, Piro R, Bardelli R, Rebelo PFS, Galeone C, Sgarbi G, Lococo F, Paci M, Ricchetti T, Cavuto S, Merlo DF, Tenconi S. PUREAIR protocol: randomized controlled trial of intensive pulmonary rehabilitation versus standard care in patients undergoing surgical resection for lung cancer. BMC Cancer. 2017 Jul 31;17(1):508. doi: 10.1186/s12885-017-3479-y. PMID 28760151
- [Background] Graham BL, Brusasco V, Burgos F, Cooper BG, Jensen R, Kendrick A, MacIntyre NR, Thompson BR, Wanger J. 2017 ERS/ATS standards for single-breath carbon monoxide uptake in the lung. Eur Respir J. 2017 Jan 3;49(1):1600016. doi: 10.1183/13993003.00016-2016. Print 2017 Jan. PMID 28049168
- [Background] Hill K, Jenkins SC, Cecins N, Philippe DL, Hillman DR, Eastwood PR. Estimating maximum work rate during incremental cycle ergometry testing from six-minute walk distance in patients with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2008 Sep;89(9):1782-7. doi: 10.1016/j.apmr.2008.01.020. PMID 18760164
- [Background] Hnizdo E, Singh T, Churchyard G. Chronic pulmonary function impairment caused by initial and recurrent pulmonary tuberculosis following treatment. Thorax. 2000 Jan;55(1):32-8. doi: 10.1136/thorax.55.1.32. PMID 10607799
- [Background] Hulya S, Naz I, Karadeniz G, Erkan S. Clinical effects of TB sequelae in patients with COPD. Int J Tuberc Lung Dis. 2022 Apr 1;26(4):363-368. doi: 10.5588/ijtld.21.0419. PMID 35351242
- [Background] Isaakidis P, Rangan S, Pradhan A, Ladomirska J, Reid T, Kielmann K. 'I cry every day': experiences of patients co-infected with HIV and multidrug-resistant tuberculosis. Trop Med Int Health. 2013 Sep;18(9):1128-1133. doi: 10.1111/tmi.12146. Epub 2013 Jul 10. PMID 23837468
- [Background] Ivanova O, Hoffmann VS, Lange C, Hoelscher M, Rachow A. Post-tuberculosis lung impairment: systematic review and meta-analysis of spirometry data from 14 621 people. Eur Respir Rev. 2023 Apr 19;32(168):220221. doi: 10.1183/16000617.0221-2022. Print 2023 Jun 30. PMID 37076175
- [Background] Khosa C, Bhatt N, Massango I, Azam K, Saathoff E, Bakuli A, Riess F, Ivanova O, Hoelscher M, Rachow A. Development of chronic lung impairment in Mozambican TB patients and associated risks. BMC Pulm Med. 2020 May 7;20(1):127. doi: 10.1186/s12890-020-1167-1. PMID 32381002
- [Background] Kosko B. Fuzzy Engineering. New Jersey: Prentice-Hall; 1997
- [Background] Lima TRL, Kasuki L, Gadelha M, Lopes AJ. Physical exercise improves functional capacity and quality of life in patients with acromegaly: a 12-week follow-up study. Endocrine. 2019 Nov;66(2):301-309. doi: 10.1007/s12020-019-02011-x. Epub 2019 Jul 17. PMID 31317523
- [Background] Lonnroth K, Migliori GB, Abubakar I, D'Ambrosio L, de Vries G, Diel R, Douglas P, Falzon D, Gaudreau MA, Goletti D, Gonzalez Ochoa ER, LoBue P, Matteelli A, Njoo H, Solovic I, Story A, Tayeb T, van der Werf MJ, Weil D, Zellweger JP, Abdel Aziz M, Al Lawati MR, Aliberti S, Arrazola de Onate W, Barreira D, Bhatia V, Blasi F, Bloom A, Bruchfeld J, Castelli F, Centis R, Chemtob D, Cirillo DM, Colorado A, Dadu A, Dahle UR, De Paoli L, Dias HM, Duarte R, Fattorini L, Gaga M, Getahun H, Glaziou P, Goguadze L, Del Granado M, Haas W, Jarvinen A, Kwon GY, Mosca D, Nahid P, Nishikiori N, Noguer I, O'Donnell J, Pace-Asciak A, Pompa MG, Popescu GG, Robalo Cordeiro C, Ronning K, Ruhwald M, Sculier JP, Simunovic A, Smith-Palmer A, Sotgiu G, Sulis G, Torres-Duque CA, Umeki K, Uplekar M, van Weezenbeek C, Vasankari T, Vitillo RJ, Voniatis C, Wanlin M, Raviglione MC. Towards tuberculosis elimination: an action framework for low-incidence countries. Eur Respir J. 2015 Apr;45(4):928-52. doi: 10.1183/09031936.00214014. PMID 25792630
- [Background] Lopes AJ, de Menezes SL, Dias CM, de Oliveira JF, Mainenti MR, Guimaraes FS. Comparison between cardiopulmonary exercise testing parameters and computed tomography findings in patients with thoracic sarcoidosis. Lung. 2011 Oct;189(5):425-31. doi: 10.1007/s00408-011-9316-1. Epub 2011 Aug 20. PMID 21858420
- [Background] Lopes AJ, Capone D, Mogami R, Lanzillotti RS, Melo PL, Jansen JM. Severity classification for idiopathic pulmonary fibrosis by using fuzzy logic. Clinics (Sao Paulo). 2011;66(6):1015-9. doi: 10.1590/s1807-59322011000600016. PMID 21808868
- [Background] Meesad P, Yen GG. Accuracy, comprehensibility and completeness evaluation of a fuzzy expert system. IJUFKS 2003; 11(4): 445-466.
- [Background] Meghji J, Lesosky M, Joekes E, Banda P, Rylance J, Gordon S, Jacob J, Zonderland H, MacPherson P, Corbett EL, Mortimer K, Squire SB. Patient outcomes associated with post-tuberculosis lung damage in Malawi: a prospective cohort study. Thorax. 2020 Mar;75(3):269-278. doi: 10.1136/thoraxjnl-2019-213808. Epub 2020 Feb 26. PMID 32102951
- [Background] Menzies NA, Quaife M, Allwood BW, Byrne AL, Coussens AK, Harries AD, Marx FM, Meghji J, Pedrazzoli D, Salomon JA, Sweeney S, van Kampen SC, Wallis RS, Houben RMGJ, Cohen T. Lifetime burden of disease due to incident tuberculosis: a global reappraisal including post-tuberculosis sequelae. Lancet Glob Health. 2021 Dec;9(12):e1679-e1687. doi: 10.1016/S2214-109X(21)00367-3. PMID 34798027
- [Background] Mpagama SG, Msaji KS, Kaswaga O, Zurba LJ, Mbelele PM, Allwood BW, Ngungwa BS, Kisonga RM, Lesosky M, Rylance J, Mortimer K. The burden and determinants of post-TB lung disease. Int J Tuberc Lung Dis. 2021 Oct 1;25(10):846-853. doi: 10.5588/ijtld.21.0278. PMID 34615582
- [Background] Migliori GB, Marx FM, Ambrosino N, Zampogna E, Schaaf HS, van der Zalm MM, Allwood B, Byrne AL, Mortimer K, Wallis RS, Fox GJ, Leung CC, Chakaya JM, Seaworth B, Rachow A, Marais BJ, Furin J, Akkerman OW, Al Yaquobi F, Amaral AFS, Borisov S, Caminero JA, Carvalho ACC, Chesov D, Codecasa LR, Teixeira RC, Dalcolmo MP, Datta S, Dinh-Xuan AT, Duarte R, Evans CA, Garcia-Garcia JM, Gunther G, Hoddinott G, Huddart S, Ivanova O, Laniado-Laborin R, Manga S, Manika K, Mariandyshev A, Mello FCQ, Mpagama SG, Munoz-Torrico M, Nahid P, Ong CWM, Palmero DJ, Piubello A, Pontali E, Silva DR, Singla R, Spanevello A, Tiberi S, Udwadia ZF, Vitacca M, Centis R, D Ambrosio L, Sotgiu G, Lange C, Visca D. Clinical standards for the assessment, management and rehabilitation of post-TB lung disease. Int J Tuberc Lung Dis. 2021 Oct 1;25(10):797-813. doi: 10.5588/ijtld.21.0425. PMID 34615577
- [Background] Migliori GB, Caminero Luna J, Kurhasani X, van den Boom M, Visca D, D'Ambrosio L, Centis R, Tiberi S. History of prevention, diagnosis, treatment and rehabilitation of pulmonary sequelae of tuberculosis. Presse Med. 2022 Sep;51(3):104112. doi: 10.1016/j.lpm.2022.104112. Epub 2022 Feb 4. PMID 35124102
- [Background] Miyamoto ST. Exercício aeróbico na síndrome de Sjogren primária: estudo controlado e randomizado. Tese de Doutorado. Universidade Federal de São Paulo. São Paulo: UNIFESP, 2016.
- [Background] Monteiro F, Ponce DA, Silva H, Carrilho AF, Pitta F. Validity and Reproducibility of the Glittre ADL-Test in Obese and Post-Bariatric Surgery Patients. Obes Surg. 2017 Jan;27(1):110-114. doi: 10.1007/s11695-016-2244-7. PMID 27317008
- [Background] Munoz-Torrico M, Rendon A, Centis R, D'Ambrosio L, Fuentes Z, Torres-Duque C, Mello F, Dalcolmo M, Perez-Padilla R, Spanevello A, Migliori GB. Is there a rationale for pulmonary rehabilitation following successful chemotherapy for tuberculosis? J Bras Pneumol. 2016 Sep-Oct;42(5):374-385. doi: 10.1590/S1806-37562016000000226. PMID 27812638
- [Background] Munoz-Torrico M, Cid-Juarez S, Gochicoa-Rangel L, Torre-Bouscolet L, Salazar-Lezama MA, Villarreal-Velarde H, Perez-Padilla R, Visca D, Centis R, D'Ambrosio L, Spanevello A, Saderi L, Sotgiu G, Migliori GB. Functional impact of sequelae in drug-susceptible and multidrug-resistant tuberculosis. Int J Tuberc Lung Dis. 2020 Jul 1;24(7):700-705. doi: 10.5588/ijtld.19.0809. PMID 32718403
- [Background] Muniyandi M, Rajeswari R, Balasubramanian R, Nirupa C, Gopi PG, Jaggarajamma K, Sheela F, Narayanan PR. Evaluation of post-treatment health-related quality of life (HRQoL) among tuberculosis patients. Int J Tuberc Lung Dis. 2007 Aug;11(8):887-92. PMID 17705955
- [Background] Neder JA, Andreoni S, Castelo-Filho A, Nery LE. Reference values for lung function tests. I. Static volumes. Braz J Med Biol Res. 1999 Jun;32(6):703-17. doi: 10.1590/s0100-879x1999000600006. PMID 10412549
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] Neder JA, Andreoni S, Peres C, Nery LE. Reference values for lung function tests. III. Carbon monoxide diffusing capacity (transfer factor). Braz J Med Biol Res. 1999 Jun;32(6):729-37. doi: 10.1590/s0100-879x1999000600008. PMID 10412551
- [Background] Nightingale R, Carlin F, Meghji J, McMullen K, Evans D, van der Zalm MM, Anthony MG, Bittencourt M, Byrne A, du Preez K, Coetzee M, Feris C, Goussard P, Hirasen K, Bouwer J, Hoddinott G, Huaman MA, Inglis-Jassiem G, Ivanova O, Karmadwala F, Schaaf HS, Schoeman I, Seddon JA, Sineke T, Solomons R, Thiart M, van Toorn R, Fujiwara PI, Romanowski K, Marais S, Hesseling AC, Johnston J, Allwood B, Muhwa JC, Mortimer K. Post-TB health and wellbeing. Int J Tuberc Lung Dis. 2023 Apr 1;27(4):248-283. doi: 10.5588/ijtld.22.0514. PMID 37035971
- [Background] Nonato CP, Azevedo BLPA, Oliveira JGM, Gardel DG, de Souza DCN, Lopes AJ. The Glittre Activities of Daily Living Test in women with scleroderma and its relation to hand function and physical capacity. Clin Biomech (Bristol). 2020 Mar;73:71-77. doi: 10.1016/j.clinbiomech.2020.01.008. Epub 2020 Jan 11. PMID 31951978
- [Background] Oostveen E, Boda K, van der Grinten CP, James AL, Young S, Nieland H, Hantos Z. Respiratory impedance in healthy subjects: baseline values and bronchodilator response. Eur Respir J. 2013 Dec;42(6):1513-23. doi: 10.1183/09031936.00126212. Epub 2013 Apr 18. PMID 23598954
- [Background] Pasipanodya JG, Miller TL, Vecino M, Munguia G, Bae S, Drewyer G, Weis SE. Using the St. George respiratory questionnaire to ascertain health quality in persons with treated pulmonary tuberculosis. Chest. 2007 Nov;132(5):1591-8. doi: 10.1378/chest.07-0755. Epub 2007 Sep 21. PMID 17890471
- [Background] Pereira CAC. Espirometria. J Bras Pneumol. 2002; 28(Supl. 3): 1-82.
- [Background] Pereira CAC, Moreira MAF. Pletismografia: resistência das vias aéreas. J Bras Pneumol. 2002; 28(3): 139-150.
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] Quaife M, Houben RMGJ, Allwood B, Cohen T, Coussens AK, Harries AD, van Kampen S, Marx FM, Sweeney S, Wallis RS, Menzies NA. Post-tuberculosis mortality and morbidity: valuing the hidden epidemic. Lancet Respir Med. 2020 Apr;8(4):332-333. doi: 10.1016/S2213-2600(20)30039-4. Epub 2020 Feb 10. No abstract available. PMID 32057300
- [Background] Ravimohan S, Kornfeld H, Weissman D, Bisson GP. Tuberculosis and lung damage: from epidemiology to pathophysiology. Eur Respir Rev. 2018 Feb 28;27(147):170077. doi: 10.1183/16000617.0077-2017. Print 2018 Mar 31. PMID 29491034
- [Background] Reis CMD, Karloh M, Fonseca FR, Biscaro RRM, Mazo GZ, Mayer AF. Functional capacity measurement: reference equations for the Glittre Activities of Daily Living test. J Bras Pneumol. 2018 Sep-Oct;44(5):370-377. doi: 10.1590/S1806-37562017000000118. Epub 2018 Jul 16. PMID 30020345
- [Background] Ross TJ. Fuzzy Logic with Engineering Applications. New York: McGraw-Hill; 1995.
- [Background] Ryu YJ, Lee JH, Chun EM, Chang JH, Shim SS. Clinical outcomes and prognostic factors in patients with tuberculous destroyed lung. Int J Tuberc Lung Dis. 2011 Feb;15(2):246-50, i. PMID 21219689
- [Background] Secretaria de Vigilância em Saúde Ministério da Saúde. Boletim Epidemiológico de Tuberculose. Número Especial -. Março 2022. Brasília: 2022. https://www.gov.br/saude/pt-br/centrais-de-conteudo/publicacoes/boletins/epidemiologicos/especiais/2022/.
- [Background] Selvaraju S, Thiruvengadam K, Watson B, Thirumalai N, Malaisamy M, Vedachalam C, Swaminathan S, Padmapriyadarsini C. Long-term Survival of Treated Tuberculosis Patients in Comparison to a General Population In South India: A Matched Cohort Study. Int J Infect Dis. 2021 Sep;110:385-393. doi: 10.1016/j.ijid.2021.07.067. Epub 2021 Jul 29. PMID 34333118
- [Background] Silva DR, Freitas AA, Guimaraes AR, D'Ambrosio L, Centis R, Munoz-Torrico M, Visca D, Migliori GB. Post-tuberculosis lung disease: a comparison of Brazilian, Italian, and Mexican cohorts. J Bras Pneumol. 2022 May 13;48(2):e20210515. doi: 10.36416/1806-3756/e20210515. eCollection 2022. PMID 35584466
- [Background] Silva DR, Gazzana MB, Barreto SS, Knorst MM. Idiopathic pulmonary fibrosis and emphysema in smokers. J Bras Pneumol. 2008 Oct;34(10):779-86. doi: 10.1590/s1806-37132008001000005. English, Portuguese. PMID 19009210
- [Background] Skumlien S, Hagelund T, Bjortuft O, Ryg MS. A field test of functional status as performance of activities of daily living in COPD patients. Respir Med. 2006 Feb;100(2):316-23. doi: 10.1016/j.rmed.2005.04.022. Epub 2005 Jun 6. PMID 15941658
- [Background] Tenconi S, Mainini C, Rapicetta C, Braglia L, Galeone C, Cavuto S, Merlo DF, Costi S, Paci M, Piro R, Fugazzaro S. Rehabilitation for lung cancer patients undergoing surgery: results of the PUREAIR randomized trial. Eur J Phys Rehabil Med. 2021 Dec;57(6):1002-1011. doi: 10.23736/S1973-9087.21.06789-7. Epub 2021 May 27. PMID 34042410
- [Background] Caglar Tosun BN, Zeren M, Barlik M, Demir E, Gulen F. Investigation of dynamic hyperinflation and its relationship with exercise capacity in children with bronchiectasis. Pediatr Pulmonol. 2022 Sep;57(9):2218-2226. doi: 10.1002/ppul.26028. Epub 2022 Jun 14. PMID 35666051
- [Background] Vashakidze SA, Kempker JA, Jakobia NA, Gogishvili SG, Nikolaishvili KA, Goginashvili LM, Magee MJ, Kempker RR. Pulmonary function and respiratory health after successful treatment of drug-resistant tuberculosis. Int J Infect Dis. 2019 May;82:66-72. doi: 10.1016/j.ijid.2019.02.039. Epub 2019 Mar 5. PMID 30844519
- [Background] Visca D, Centis R, Munoz-Torrico M, Pontali E. Post-tuberculosis sequelae: the need to look beyond treatment outcome. Int J Tuberc Lung Dis. 2020 Aug 1;24(8):761-762. doi: 10.5588/ijtld.20.0488. No abstract available. PMID 32912378
- [Background] Visca D, Zampogna E, Sotgiu G, Centis R, Saderi L, D'Ambrosio L, Pegoraro V, Pignatti P, Munoz-Torrico M, Migliori GB, Spanevello A. Pulmonary rehabilitation is effective in patients with tuberculosis pulmonary sequelae. Eur Respir J. 2019 Mar 14;53(3):1802184. doi: 10.1183/13993003.02184-2018. Print 2019 Mar. No abstract available. PMID 30872556
- [Background] Wang J, Xiong K, Zhao S, Zhang C, Zhang J, Xu L, Ma A. Long-Term Effects of Multi-Drug-Resistant Tuberculosis Treatment on Gut Microbiota and Its Health Consequences. Front Microbiol. 2020 Jan 30;11:53. doi: 10.3389/fmicb.2020.00053. eCollection 2020. PMID 32082283
- [Background] World Health Organization. Global tuberculosis report 2021]. Geneva: WHO; 2021. Global Tuberculosis Report 2021. Disponível em: https://www.who.int/publications/i/item/9789240037021.
- [Background] World Health Organization. Global Tuberculosis Report 2022. Geneva: WHO; c2022. Disponível em: https://www.who.int/teams/global-tuberculosis-programme/tbreports/global-tuberculosis-report-2022.
- [Derived] Souza AMLR, Silva DLOD, Silva MMD, Silva LLD, Silva UDPVD, Beserra ADS, Freitas YO, Ferreira IDN, Lopes AJ. Peripheral Muscle Strength and Pulmonary Function Negatively Impact Functional Capacity in Patients With Post-Tuberculosis Lung Disease: A Cross-Sectional Study. Physiother Res Int. 2025 Oct;30(4):e70115. doi: 10.1002/pri.70115. PMID 41035122